CLINICAL TRIAL: NCT05306171
Title: Effects of Online Training on Self-esteem and Occupational Stress of Healthcare Professionals: a Possible Strategy for Prevention of Burnout Syndrome.
Brief Title: Online Training for Healthcare Professionals: a Possible Strategy for Prevention of Burnout
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Carlos Vicente Serrano Jr, Director, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SDC 4734/18/085
Record Dates: First submitted 2022-03-10; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Burnout
Keywords: Burnout Syndrome; Self Esteem; Occupational Stress; Online Training; Health Professionals
MeSH Terms: conditions — Burnout, Psychological; Occupational Stress | interventions — Health Personnel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (I) (Experimental): Online training for healthcare professionals which will follow a protocol made especially for this research. The online training is composed by 4 modules and each module has 3 meetings. Each meeting has 35 minutes long.
  Interventions: Behavioral: Online training for healthcare professionals
- Control group (C) (No Intervention): No intervention. The control group will receive the intervention after study is completed.

INTERVENTIONS:
Behavioral: Online training for healthcare professionals — The online training (4 modules) will use the technique of hybrid learning, combining meetings that will require the presence of participants and mediator at the same time and platform (live) with recorded meetings (interviews with experts) that will be watched by the participants at any time (from a distance).
  Module 1: Self Care; Module 2: Stress and anxiety management; Module 3: Relationships; Module 4: Communication.
  Arms: Intervention group (I)

SUMMARY:
This study aims to evaluate the effects of online training on self-esteem and occupational stress of healthcare professionals, in order to evaluate the potential of this intervention as a preventive measure to Burnout syndrome. The study will be developed in three phases,the first being the period of one week before the intervention(t0), when instruments will be first applied.The second phase corresponds to intervention period, when the instruments will be reapplied after the second (t1), third (t2) and fourth (t3) training intervention. The third phase corresponds to the follow up (t4-t8), when all instruments used in the second phase will be reapplied in 2 months (t4), 4 months (t5), 6 months (t6), 8 months (t7) and 12 months (t8) after the end of the intervention.

The sample will consist of 100 health professionals randomized into two groups (50 in each group): intervention group (I), formed by those who will participate in the online training and control group (C), formed by those who will receive the intervention after research is finished.

The hypotheses are: the online training will have greater effect on the increase of self-esteem, and will be identified in health professionals: low levels of global self-esteem, high levels of occupational stress and average levels of burnout.

ELIGIBILITY:
Inclusion Criteria:

* Health professionals who work at University of Sao Paulo General Hospital
* Agree and sign the Inform Consent Form.

Exclusion Criteria:

* Those who, one week before training, presents anxiety and depressive symptoms (GAD ≥ 14 e/ou PHQ ≥ 14)
* in psychotherapy during data collection;
* diagnosed with Burnout syndrome.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Self esteem | Through study completion, an average of 1 year and 4 months
  Assessed by the instrument Rosenberg Self Esteem Scale(RSES)
Occupational Stress | Through study completion, an average of 1 year and 4 months
  Assessed by the instrument Stress Questionnaire for Health Professionals (SQHP)
Burnout | Through study completion, an average of 1 year and 4 months
  Assessed by the instrument Copenhagen Burnout Inventory(CBI)

SECONDARY OUTCOMES:
Anxiety | Through study completion, an average of 1 year and 4 months
  Assessed by the instrument Generalized Anxiety Disorder-7 (GAD-7)
Depression | Through study completion, an average of 1 year and 4 months
  Assessed by the instrument Patient Health Questionnaire - 9 (PHQ-9)
Covid-19 impact | Through study completion, an average of 1 year and 4 months
  Assessed by the instrument Impact of Event Scale - Revised (IES -Rs)
Improvement in general health after entering the study. | Through study completion, an average of 1 year and 2 months
  Assessed by the instrument Patient Global Improvement Change Scale (PGIC)

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia Perniciotti Almeida Costa, Phd student, Principal Investigator — University of Sao Paulo Medical School
Locations (1):
- Heart Institute of the Hospital das Clínicas, University of São Paulo Medical School, São Paulo, Brazil